CLINICAL TRIAL: NCT03563963
Title: Evaluating Ropivacaine and Lidocaine in the Endotracheal Tube Cuff on Post-Operative Sore Throat Incidence and Severity - A Randomized Clinical Trial
Brief Title: Ropivacaine vs Lidocaine in the Endotracheal Tube Cuff on Post-Operative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bio 18-09
Record Dates: First submitted 2018-05-22; First posted 2018-06-20 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pharyngitis; Lidocaine; Ropivacaine; Intubation, Intratracheal; Post-operative Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Ropivacaine; Lidocaine; Air

STUDY DESIGN:
Intervention Model Description: The two intervention groups will be: 1) lidocaine 2% in the ETT cuff and 2) ropivacaine 0.5%in the ETT cuff. The control group will be air in the ETT cuff.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesia provider will be blinded to the intervention group allocation as the two solutions are clear, however they will not be blinded if their patient is in the control group. All patients will be anesthetized when the medium is placed in the ETT, thus patients will be blinded. The primary investigator will be blinded. The resident researcher who will be the outcome assessor will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine 2% in Endotracheal Tube cuff (Active Comparator): Lidocaine 2% will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Interventions: Drug: Lidocaine 2% Preservative-Free Injectable Solution
- Ropivacaine 0.5% Endotracheal Tube cuff (Experimental): Ropivacaine 0.5% will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- Air in the Endotracheal Tube cuff (Active Comparator): Air will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Interventions: Other: Air

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Ropivacaine 0.5% will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Arms: Ropivacaine 0.5% Endotracheal Tube cuff
Drug: Lidocaine 2% Preservative-Free Injectable Solution — Lidocaine 2% will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Arms: Lidocaine 2% in Endotracheal Tube cuff
Other: Air — Air will used to inflate the endotracheal tube cuff using the stethoscope guided inflation technique described by Kumar and Hirsch (2). The anesthesiologist will documented the volume in millilitres instilled into the cuff to create a seal. Once a seal was created the anesthesiologist will documented the ETT cuff pressure. If an endotracheal cuff leak occurred during the surgical procedure, the randomized solution was used to inflate the cuff.
  Arms: Air in the Endotracheal Tube cuff

SUMMARY:
In elective gynecology and general surgery patients age 18 and over requiring endotracheal tube (ETT) intubation, what is the efficacy of ropivacaine 0.5% vs. lidocaine 2% as the medium to inflate the ETT cuff, compared to the standard of air, in reducing the incidence and severity of POST on post-op day one?

DETAILED DESCRIPTION:
We plan a randomized clinical trial comparing postoperative sore throat between three groups: 1) ETT cuff inflated with ropivacaine, 2) ETT cuff inflated with lidocaine, and 3) ETT cuff inflated with air (standard care).

The Saskatoon Health Region has on average 24 elective operating rooms in use every weekday, with tracheal intubation being a common intervention in patients coming for surgery. To aid with homogeneity, only ASA 1-3 gynecology and general surgery patients who require endotracheal intubation with major surgery criteria will be recruited. The criteria for major surgery will be defined as those that require hospitalization for more than one day.(1) Patients under the age of 18 and those with pre-operative sore throat will be excluded. In the pre-operative holding area, the anesthesia provider will explain the risk of anesthesia. Oral and written consent will be obtained after the anesthesia provider (staff or resident) has explained the risk and benefits of the research project. After informed consent has been received the patients will be randomized to one of the two intervention groups or to the control using computer-generalized random sequence. The anesthetic provided will be chosen based on clinical grounds as per the anesthesiologist's discretion. The following will be documented by the anesthesiologist: if an oral airway was used at any time, size of endotracheal tube, number of intubation attempts, the Cormack-Lehane intubation grade, the number of intubation attempts required to be successful, and if a stylet was required to secure the ETT. The ETT cuff will be inflated with either lidocaine 2%, ropivacaine 0.5%, or air. To inflate the cuff, the stethoscope guided inflation technique will be used.(2) For all groups, the anesthetist will document the volume in milliliters instilled into the cuff. Nitrous oxide will not be used at any time during the anesthetic, as nitrous oxide is associated with an increase of the ETT cuff pressure and thus potential for mucosal damage.(3) The anesthesia provider will not be blinded to the interventions. All patients will be anesthetized when the medium is placed in the ETT, thus patients will be blinded. Gentle suctioning of the oropharynx may be administered at the end of the surgery.

Documentation will be made if patients are smokers or have hyperactive airway disease (ex. asthma, COPD, or URTI in the last 4 weeks). In addition, age, sex, ASA status, duration of intubation and type of surgery will be documented. The anesthesia provider will make note of the incidence of coughing prior to extubation as mild (<5 coughs), moderate (5-10 coughs), or severe (>10 coughs); with cough defined as the sudden expelling of air from the lungs with a loud noise. Prior to discharge from the post anesthetic care unit (PACU), the resident researcher who is blinded to patient allocation will assess for the presence of sore throat (defined as pain in the throat) with a "yes" or "no" evaluation. If patients report yes, then they will be report the severity using the Numerical Rating Scale (NRS) of 0-10.(4) Surgical site pain will be assessed using the NRS of 0-10. The following will also be noted in PACU: the presence of dysphagia (defined as difficulty in swallowing), and hoarseness or dysphonia (defined as a rough or harsh voice pattern) by a "yes" or "no" evaluation. The time spent in PACU will also be recorded.

The resident researcher will perform bed side evaluation of all participants on post-op day one for the presence of sore throat with a "yes" or "no" evaluation. If patients indicate "yes", then the severity will be reported using the NRS. To ensure surgical pain is not distracting patients, the research will also assess surgical pain using the NRS. The presence of dysphagia and hoarseness or dysphonia will be assessed by a "yes" or "no" evaluation. Finally, patient satisfaction with their anesthesia will be assessed on post-operative day 1 with a 5-point Likert scale with the following categories: very satisfied, satisfied, neither, dissatisfied, or very dissatisfied. If a patient is discharged home on post-op day one prior to the resident researcher performing the bed side evaluation, the patient will be contacted by phone using the phone number proved at the time of hospital registration.

The sample size for the study is based on studies included in the meta-analysis by Lam et al. (5) The sample size required to provide a 80% power for a 0.05 significance level between the three groups is 14 per group, but 20 per group will be recruitment to account for patient drop-out.

The data will be collected by the resident researcher. Statistical analysis will be completed by a statistician within the anesthesia department. The outcomes of POST, surgery pain, dysphagia and hoarseness in the PACU and POD1, as well as the outcomes cough and cuff-pressure, will be analyzed using Pearson chi-square. Fisher's Exact test will be used where cell count of a variable is less than five. Effect size for the categorical primary and secondary outcomes will be calculated using Cramer's V and the effect size for the continuous secondary outcomes will be calculated using Eta squared (ƞ2) for Kruskal Wallis-H. If continuous variable score do not follow normal distributions we will compare the continuous variables for treatment groups (air, ropivacaine and lidocaine) using the Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecology and general surgery patients
* Age 18 or older
* Must be coming for a surgical procedure that requires having a general -anesthetic requiring endotracheal intubation
* Must be admitted to hospital for more than one day
* ASA class 1-3 inclusive

Exclusion Criteria:

* Pre-operative sore throat the day of of recruitment
* Upper respiratory tract infection in the previous 4 weeks
* Intra-operative use of transesophageal echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Post-operative sore throat | Post-operative day one
  Using Numerical Rating Scale of 0-10

SECONDARY OUTCOMES:
Incidence of cough at extubation | From time of surgery closure plus one hour
  Mild (<5 coughs), moderate (5-10 coughs), or severe (>10 coughs)
Post-operative sore throat | Prior to leaving post anesthetic care unit plus two hours
  Using Numerical Rating Scale of 0-10
Time spent in post anesthetic care unit (PACU) | Surgical day zero
  From time entered PACU until criteria met to be discharged from PACU
Dysphagia | Once criteria met to be discharged from the post anesthetic care unit plus two hours, and on post operative day one up to 36 hours post-op
  Incidence of dysphagia (defined as difficulty in swallowing)
Patient satisfaction | Post-operative day one
  Using a 5-point Likert scale with the following categories: very satisfied, satisfied, neither, dissatisfied, or very dissatisfied
Surgical site pain score | Once criteria met to be discharged from the post anesthetic care unit plus two hours, and and on post operative day one up to 36 hours post-op
  Using Numerical Rating Scale of 0-10
Dysphonia | Once criteria met to be discharged from the post anesthetic care unit plus two hours, and and on post operative day one up to 36 hours post-op
  Incidence of dysphonia (defined as a rough or harsh voice pattern)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, MD, FRCPC, Principal Investigator — Department of Anesthesiology, Perioperative Medicine and Pain Management, University of Saskatchewan
Locations (2):
- Canada (2):
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Saskatoon City Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang YW, Chou YC, Yeh CC, Hu CJ, Hung CJ, Lin CS, Chen TL, Liao CC. Outcomes after major surgery in patients with myasthenia gravis: A nationwide matched cohort study. PLoS One. 2017 Jun 30;12(6):e0180433. doi: 10.1371/journal.pone.0180433. eCollection 2017. PMID 28666024
- [Background] Kumar RD, Hirsch NP. Clinical evaluation of stethoscope-guided inflation of tracheal tube cuffs. Anaesthesia. 2011 Nov;66(11):1012-6. doi: 10.1111/j.1365-2044.2011.06853.x. Epub 2011 Aug 18. PMID 21851343
- [Background] Navarro RM, Baughman VL. Lidocaine in the endotracheal tube cuff reduces postoperative sore throat. J Clin Anesth. 1997 Aug;9(5):394-7. doi: 10.1016/s0952-8180(97)00068-8. PMID 9257206
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Lam F, Lin YC, Tsai HC, Chen TL, Tam KW, Chen CY. Effect of Intracuff Lidocaine on Postoperative Sore Throat and the Emergence Phenomenon: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Aug 19;10(8):e0136184. doi: 10.1371/journal.pone.0136184. eCollection 2015. PMID 26288276